| 'The Effect Of Nutrition And Fluid Intake İn The First Stage Of Labor On Maternal And |
|---|
| Fetal Outcomes' |
| NCT Number: |
| 22.03.2022 |

Birth is a process that requires large amounts of energy. As a result of skeletal and smooth muscle contractions at birth, the body's basal metabolic rate, energy requirement, hydration requirement, and insensible fluid loss are significantly increased. Information regarding the safety and effectiveness of increased hydration during labor is still controversial. There has yet to be a consensus on whether this hydration should be given with intravenous solutions or orally. The study aims to determine the effect of fluid intake in labor on the delivery process, maternal-fetal outcomes.

## Inclusion Criteria:

- Volunteer to participate in the research
- Agreeing to abide by the protocol
- Being able to read and write,
- Ages 18-35 years
- 37-40 Pregnancy weeks
- First pregnancy,
- Single fetus
- BMI  $\leq$  28,
- Head presentation
- Cervical dilatation of <6 cm or less (latent phase)
- Height  $\geq 1.50$  cm

## **Exclusion Criteria**:

- Communication barriers (speech, hearing, mental),
- Disability (physical or mental problem, drug use),
- Chronic diseases (hypertension, diabetes, etc),
- Gastrointestinal problems before and during pregnancy
- Comply with the fluid intake protocol during labor,
- Pregnant women who are scheduled for elective cesarean section
- Pregnant women considered to be at immediate cesarean risks, such as diabetic pregnant women with cephalopelvic incompatibility, multiple pregnancies, preeclampsia, and macrosomic fetus

## Methods of Study:

The study was planned as a randomized controlled experimental study to evaluate the effect of fluid intake during labor on mothers and babies. Location and Characteristics of the Research: The research will be conducted in the delivery room of Sakarya Training and Research Hospital. Population and Sample of the Study: The research will consist of pregnant women who apply to Sakarya Training and Research Hospital with signs of the onset of labor and will have an expected vaginal delivery in the delivery room. Annually, 7000-8000 women give birth in the hospital, and approximately 50% have an expected vaginal delivery. All pregnant women who met the sampling criteria and volunteered to participate during the study's implementation will be included. The research will be carried out in 3 groups experimental and control groups. The study will be conducted with a total of 90 pregnant women, 30 of whom are in each group. Outcomes: During the research, the week of pregnancy, examination findings (cervical dilation and effacement), duration of the latent phase of labor, and active phase of labor (time from 6 cm cervical dilation to the birth), oxytocin need, delivery type, postpartum bleeding, fetal weight, APGAR scores, whether the newborn is admitted to the intensive care unit, maternal pain visual analog scale (VAS) scores will be recorded. Fluid monitoring will be done separately for all groups. After labor, 100 ml of fruit juice and water will be taken orally, and iv hydration will be calculated in the delivery room midwife records. VAS scores determine the pain levels of women in the experimental and control groups in the latent phase of labor (cervical dilatation 3-4 cm), the active phase (cervical dilatation 8-10 cm), and the early postpartum period (within the first 15 minutes). It will be applied three times in total. The study will be conducted from the latent phase of labor to birth.